CLINICAL TRIAL: NCT05302752
Title: Quantification and Repeatability of Responses to Rapid Bilateral Magnetic Stimulation of the Phrenic Nerves
Brief Title: Quantification and Repeatability of Magnetic Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REMEX-WP1
Record Dates: First submitted 2022-03-18; First posted 2022-03-31 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bilateral rapid magnetic stimulation of the phrenic nerves (Experimental): Each participant will be tested on three different days with optimal settings for bilateral rapid magnetic stimulation of the phrenic nerves established on visit 1 and then repeated on visits 2 and 3.
  Interventions: Other: Magnetic phrenic nerve stimulation

INTERVENTIONS:
Other: Magnetic phrenic nerve stimulation — The intervention consists of bilateral rapid magnetic phrenic nerve stimulation on the neck using different stimulation intensities.
  On one visit, the effect of increasing chest wall stiffness and respiratory muscle work by adding incrementally small weights to the chest/abdomen will be investigated.

SUMMARY:
In this project the quantification and the repeatability of responses to rapid bilateral magnetic stimulation of the phrenic nerves will be investigated in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* normal lung function
* body mass index: 18.5-29.9 kg/m2
* able to communicate in english
* willing to adhere to study rules

Exclusion Criteria:

* acute illness or chronic conditions of the gastrointestinal tract, and health conditions affecting metabolism, the cardiovascular or the respiratory system, or sleep
* intake of medications affecting metabolism, the cardiovascular, the neuromuscular or the respiratory system, or sleep
* any metal or electronics inside of the body
* presence of cardiac pacemaker, implanted defibrillators or implanted neurostimulators
* history of seizures or epilepsy
* tatoos on the stimulation sites
* previous enrolment in this study
* for women: pregnancy, breastfeeding, or intention to become pregnant during the study

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Diaphragm contractility | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec
  Transdiaphragmatic pressure changes, i.e. changes in esophageal and gastric pressures, will be measured by a pressure transducer connected to balloon-catheters.

OTHER OUTCOMES:
Changes in airflow | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Flow will be recorded by a pneumotachometer and averaged over breaths.
Changes in chest and abdominal movements | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Chest and abdominal movements will be assessed using respiratory belt strain transducers.
Changes in costal diaphragm activity | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Costal diaphragm activity will be continuously recorded via a wireless surface electromyography system.
Head, shoulder and arm accelerations | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Head, shoulder and arm movements will be recorded using wireless acceleration sensors attached to the head and arms.
Body movement | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Overall body movement incl. head, shoulder and arm movements will be recorded using a video camera.
Changes in skin conductance | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Skin conductance (μS) will be continuously recorded with electrodes worn on two fingers.
Changes in heart rate | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Heart rate will will be continuously recorded beat by beat (1/min) with electrodes on both wrists and one ankle.
Changes in blood pressure | Continuously measured from 10 sec before until 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Systolic and diastolic blood pressure (mmHg) will be continuously recorded using a non-invasive device.
Perception of pain, paresthesia and discomfort | Assessed 10 sec after each stimulation. One stimulation lasts for approx. 1 sec.
  Participant subject perception of pain, paresthesia and discomfort will be evaluated with 0-to-10-point scale, with 0 = no pain/paresthesia/discomfort and 10 = maximal pain/paresthesia/discomfort. Higher values indicate more perception of the specified sensations.

CONTACTS AND LOCATIONS:
Overall Officials: Christina M. Spengler, Prof., Principal Investigator — ETH Zurich, Exercise Physiology Lab, Institute of Human Movement Sciences and Sport
Locations (1):
- Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No